CLINICAL TRIAL: NCT02727296
Title: Volatile Anesthetic Protection Of Renal Transplants 2
Acronym: VAPOR-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Gertrude J. Nieuwenhuijs-Moeke, MD PhD, MD PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAPOR-002
Record Dates: First submitted 2016-03-23; First posted 2016-04-04 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Delayed Graft Function; Renal Outcome After Kidney Transplantation; Acute Rejection (AR) of Transplanted Kidney; Graft Survival; Patient Survival; Postoperative Complications; Length of Hospital Stay; Primary Non Function
Keywords: anesthesiology; sevoflurane; propofol; kidney transplantation
MeSH Terms: conditions — Delayed Graft Function; Postoperative Complications | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- propofol (Active Comparator): Group 1 PROP (control): propofol: a propofol-remifentanil based general anesthesia.
  Interventions: Drug: propofol
- sevoflurane (Active Comparator): Group 2 SEVO (intervention): Sevoflurane: a sevoflurane-remifentanil based general anesthesia.
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: sevoflurane — General anesthesia with sevoflurane
  Arms: sevoflurane
Drug: propofol — General anesthesia with propofol
  Arms: propofol

SUMMARY:
To compare the effect of a sevoflurane based anesthesia versus a propofol based anesthesia on the incidence of DGF in recipients of kidneys of donation after circulatory death (DCD) and donation after brain death (DBD) donors

DETAILED DESCRIPTION:
Objective:

To compare the effect of a sevoflurane based anaesthesia versus a propofol based anaesthesia on the incidence of delayed graft function in recipients of DCD and DBD donor kidneys.

Study design:

Prospective randomized controlled European multicentre clinical trial with two parallel groups

Study population:

Patients ≥18 years scheduled for kidney transplantation with a kidney from a DBD or DCD donor

Intervention:

Patients will be included and randomised to one of the following groups:

Group 1 PROP (control): Propofol: a propofol-remifentanil based anaesthesia. Group 2 SEVO (intervention): Sevoflurane: a sevoflurane-remifentanil based anaesthesia.

Main study parameters:

Primary outcome: The two co-primary endpoints are the incidence of DGF and one-year acute rejection in recipients of DCD and DBD donor kidneys. DGF is defined as need for dialysis within the first week after transplantation, excluding one-time dialysis for hyperkalaemia. Acute rejection is defined by the modified BANFF 2013 classification and must be associated with decline in kidney function and treatment.

Secondary outcomes Functional delayed graft function (fDGF) is defined as the absence of a daily decrease of at least 10% in serum creatinine for at least three consecutive days; primary non function (PNF) defined as a permanent lack of function of the allograft; length of hospital stay and postoperative complications of all kind (28). Estimated glomerular filtration rate (eGFR) at one week and three and twelve months calculated with the CKD-EPI formula; measured GFR employing Iodinethalamate (Groningen), CrEDTA (Aarhus) and Iohexol (Oslo) at twelve months; readmissions at three and twelve months, graft survival and patient survival at twelve months.;

The investigators predefined four substudies being: Cardiac biomarkers in renal transplantation, Volatile vs Intravenous anaesthetic agent; Predictive value of urinary Biomarkers in a deceased donor kidney transplantation cohort to predict PNF, DGF, Acute rejection and long term graft function and outcome; Association between intraoperative haemodynamics and vasopressor use and graft outcome; Postoperative delirium, volatile vs Intravenous anaesthetic agent (Groningen, Aarhus);

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Written informed consent

Exclusion Criteria:

* high immunological risk as determined bij local practice
* Patients of the ABO-incompatible program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of delayed graft function and/or one year acute rejection | DGF: 7 days after transplantation Acute rejection: up to 1 year after transplantation
  DGF is defined as need of dialysis first 7 days after transplantation Acute rejection up to 1 year after transplantation, defined by the modified BANFF 2013 classification and must be associated with decline in kidney function and treatment.

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate (GFR) | 7 days after transplantation, 3 months after transplantation, 1 year after transplantation
  calculated with the CKD-EPI formula
incidence of primary non function (PNF) | up to 3 months after transplantation
  PNF is defined as permanent lack of function of the transplanted kidney. This kidney will not gain function after transplantation
Incidence of funactional Delayed Graft Function | 7 days after transplantation
  Absence of a daily decrease of at least 10% in serum creatinine for at least three consecutive days
Length of hospital stay | From day of transplantation until the day of discharge, assessed up to 60 days
  Days
Postoperative complications of all kind | from the day of transplantation until the day of discharge, assessed up to 60 days
hospital readmissions after transplantation | 3 months after transplantation and between 3 months and 1year after transplantation
Graft survival | up to 1 year after transplantation
All-cause mortality | up to 1 year after transplantation
  Mortality due to any cause
measured GFR employing Iodinethalamate (Groningen), CrEDTA (Aarhus) and Iohexol (Oslo) at twelve months | 1 year after transplantation
  In a subpopulation of Groningen, Aarhus, Oslo; employing Iodinethalamate (Groningen), CrEDTA (Aarhus) and Iohexol (Oslo)

OTHER OUTCOMES:
Cardiac biomarkers in renal transplantation, Volatile vs Intravenous anesthetic agent. A substudy of the VAPOR-2 study; a multicenter randomized controlled study | From enrollment to 1 year follow-up
  The aim of our study is to investigate cardiac biomarkers in kidney transplant recipients using two different anesthesia regimen and to investigate whether there is any difference in outcome. In this substudy we will investigate the levels and thresholds of cardiac biomarkers (Troponin-T and pro-BNP) at three time points (day 0, day 1 and day3) with two different anesthetic management (intravenous or inhalational), and the impact of outcome and MACE (major adverse cardiac events). The findings in this study may provide important information for the transplant team about which anesthesia is best suited for kidney transplant recipients with cardiovascular comorbidity.
Predictive value of urinary Biomarkers in a deceased donor kidney transplantation cohort to predict PNF, DGF, Acute rejection and long term graft function and outcome | from enrollement to follow-up of 1 year
  The donation and transplantation procedure is inevitably accompanied by harmful processes that impact the kidney's viability. Ischemia reperfusion injury (IRI) is one of the main harmful processes which frequently results in complications and reduced kidney function after transplantation, such as delayed graft function (DGF) or primary non-function (PNF) . It is therefore important to detect and prevent damage as a result of IRI. An improved and earlier detection of IRI-induced damage might allow therapeutic measures and improve renal function and patient outcome on a longer term. We studied several biomarkers in a living donor kidney transplantation (LDKT) cohort. We will now proceed whit analysis of the release pattern and predictive value of KIM-1, H-FABP, NAG and NGAL and novel biomarkers on short- and long-term graft outcome after deceased donor kidney transplantation
Association between intraoperative haemodynamics and graft outcome | from enrollement to 1 year follow-up
  Perioperative hemodynamic and fluid management remains one of the most debated topics in modern anesthesia, particularly in the context of kidney transplantation, where there is currently no consensus on optimal blood pressure targets. This is further complicated by the fact that the transplanted kidney is denervated, resulting in impaired autoregulation and making renal blood flow directly dependent on systemic circulation. Our objective is to identify specific intraoperative hemodynamic parameters that are associated with both short- and long-term graft outcomes. To achieve this, we will analyze continuous intraoperative hemodynamic data and assess their relationship with delayed graft function (DGF), acute rejection (AR), primary non-function (PNF), estimated glomerular filtration rate (eGFR) at 3 and 12 months, and overall graft survival.
Incidence of postoperative delirium assessed by RASS in PACU and CAM on postoperative days 1-2 between volatile vs Intravenous anaesthetic agent, A substudy of the VAPOR-2 study | From day of transplantation until 2 days postoperative
  This substudy investigates the incidence of postoperative delirium after renal transplantation in a randomized controlled trial with two groups anesthetized using either Propofol or Sevoflurane. Postoperative delirium will be screened using RASS (Richmond agitation sedation score) in the PACU and CAM (Confusion assessment method) during the first two postoperative days on the ward.
  The findings from this study will provide information about the incidence of postoperative delirium following renal transplantation. Data may provide information about differences depending on the choice of anesthetic agent - Propofol versus Sevoflurane.

CONTACTS AND LOCATIONS:
Overall Officials: Gertrude J Nieuwenhuijs-Moeke, MD, Principal Investigator — University Medical Center Groningen
Locations (5):
- Aarhus University Hospital, Aarhus, Denmark
- Netherlands (2):
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Amsterdam University Medical Center, Amsterdam
- university Hospital Oslo, Oslo, Norway
- Fundagio Puigvert, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study and primary data analysis, the dataset will be anonymized and made openly accessible through a public data repository
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study Protocol, ICF and SAP will be shared with the protocol article which will be publihed open access Upon completion of the study and primary data analysis, the dataset will be anonymized and made openly accessible through a public data repository (start date January 2027-end date to be determined)
Access Criteria: all will be open access

REFERENCES:
- [Derived] Huisman GJJ, Berger SP, Thyrrestrup PS, Hausken J, Veelo DP, Guirado L, Pol R, Jensen LL, Tonnessen TI, Bemelman FJ, Facundo C; VAPOR-2 STUDY GROUP; Tamasi K, Lunter G, Jespersen B, Leuvenink HGD, Struys MMRF, Nieuwenhuijs-Moeke GJ. Propofol-based versus sevoflurane-based anaesthesia for deceased donor kidney transplantation: the VAPOR-2 study protocol for an international multicentre randomised controlled trial. BMJ Open. 2025 Sep 2;15(9):e098965. doi: 10.1136/bmjopen-2025-098965. PMID 40897490